CLINICAL TRIAL: NCT01511965
Title: Study of Applications of Autologous Epidermal Cells in Liquid Phase in the Treatment of Vitiligo
Acronym: Viticell
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-API-01
Record Dates: First submitted 2012-01-02; First posted 2012-01-19 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Cell- and Tissue-Based Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- traitement A (Other): Lesion 1= graft and lesion 2 = UltraViolet B
  Interventions: Other: autologous (cellular therapy)
- traitement B (Other): Lesion 1 = UltraViolet B and lesion 2 = graft
  Interventions: Other: autologous (cellular therapy)

INTERVENTIONS:
Other: autologous (cellular therapy) — The skin sample, the preparation and implementation of the epidermal cells, are conducted on one day. A review of selected lesions is performed and a photograph. Second, are performed successively in a single day the collection of thin skin, preparing the cell suspension, a desepidermisation laser Erbium: YAG lesions of vitiligo to be grafted, and applicated.

SUMMARY:
Vitiligo is a depigmenting skin disease common. Vitiligo is caused by the disappearance of melanocytes in the epidermis. Vitiligo is the cause of disfigurement, psychological and social, that sounds a lot about the quality of life. Currently the standard treatment for vitiligo is ultraviolet ray (UV), but it only allows a 50% repigmentation of lesions in half of patients. The applications of autologous epidermal cells in the liquid phase is a promising new therapeutic approach of vitiligo.

The main goal of this study is to compare prospectively the repigmentation of vitiligo lesions induced by application of autologous epidermal cells in liquid phase associated with light therapy and light therapy alone.

Study's secondary goals: compare the applications of epidermal cells to phototherapy alone and phototherapy, in respect of:

* Obtain a repigmentation> 70% (threshold considered aesthetically relevant)
* The occurrence of adverse events
* Patient satisfaction regarding the efficacy and safety of treatment

DETAILED DESCRIPTION:
MAIN CRITERIA

* Rates of repigmentation of the vitiligo lesions to 12 months
* The lesions of the layers defined by the investigator to Month 0, Month 3, Month 6 and Month 12 will be analyzed by an image analysis system managed by a computer.
* Digital photos is taken in order to illustrate the quantitative results above.

SECONDARY CRITERIA

* Repigmentation> 70% of the vitiligo lesions at 12 months
* Rates of repigmentation of the vitiligo lesions at 12 months
* Side effects: the frequency, severity and time of occurrence will be reported for each treatment. Side effects are classified into grades according to World Health Organization (WHO) criteria.
* Patient satisfaction of the effectiveness and tolerance will be studied using visual analogue scales graded from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients at least 18 years
* Subjects with a stable vitiligo (no new injury or lack of expansion of existing lesions in the last 12 months), with at least two vitiligo lesions of at least 10 cm2 located in the same anatomical location, and requiring treatment with UVB phototherapy.
* Topic with vitiligo
* Subjects who agreed to have a blood research with Human immunodeficiency virus (HIV), Human T-lymphotropic virus - 1 (HTLV-1), hepatitis B, hepatitis C, and human Chorionic Gonadotropinfor (hCG) women.
* For women of childbearing age, the use of effective contraception (birth control pills or Intrauterine Device (IUD)) for the duration of the study
* Topics able to participate and to respect it.
* Topics affiliated to social security.
* Topics that have signed a written informed consent before the start of the study.

Exclusion Criteria:

* Pregnant or nursing women.
* Subjects with a history of keloid scarring.
* Subjects with a history of melanoma.
* Subjects with a photodermatitis.
* Topics taking photosensitizing treatment.
* Subjects who received treatment for vitiligo in the 4 weeks before enrollment.
* Subjects with HIV testing, hepatitis B or hepatitis C positive.
* Major Topics protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Rate of repigmentation of vitiligo lesion to 12 months | 12 months
  The lesions defined by the investigator to Month 0, Month 3, Month 6 and Month 12 will be analyzed by an image analysis system managed by a PC computer. Digital photos will be taken in order to illustrate the quantitative results above.

SECONDARY OUTCOMES:
Repigmentation> 70% of vitiligo lesion at 6 months | 6 months
Side effects | 12 months
  the frequency, severity and time of occurrence of side effects will be reported for each treatment. Side effects are classified into grades according to WHO criteria.
Patient satisfaction | 12 months
  Patient satisfaction and tolerance will be studied using visual analogue scales graded from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Bahadoran, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- service de Dermatologie - Hôpital l'Archet, Nice, France